CLINICAL TRIAL: NCT07215949
Title: Zilucoplan Treatment of Severe MG Exacerbations Leading to Hospitalization of Participants With Acetylcholine Receptor Antibody Positive gMG
Brief Title: Zilucoplan for Severe gMG Exacerbations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Miriam Freimer (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Miriam Freimer, Professor of Neurology, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0036-OSU
Record Dates: First submitted 2025-10-06; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Generalized Myasthenia Gravis (gMG)
Keywords: MG; exacerbation; zilucoplan
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilucoplan (Experimental): Subcutaneous zilucoplan
  Interventions: Drug: Zilucoplan®

INTERVENTIONS:
Drug: Zilucoplan® — Subcutaneous injections of zilucoplan will be administered daily. The dose is dependent on the body weight of the patient. Each patient will receive a kit with prefilled syringes.

SUMMARY:
This is an open-label, multicenter, interventional phase 3b study in participants with AChR+ gMG and severe exacerbation that require hospitalization. Patients will receive subcutaneous zilucoplan injections daily for 12 weeks. Participation in the study will last for approximately 18 weeks.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of subcutaneous zilucoplan in participants with AChR antibody positive gMG who experience severe exacerbations requiring hospitalization. A total of 15 patients will be enrolled in the study with treatment lasting 12 weeks. Dosing will be weight based.

Patients will be presented with the option of undergoing standard of care plasma exchange or IVIG or to participate in the research study to determine if the use of zilucoplan would rapidly alleviate the most severe symptoms of gMG (respiratory dysfunction and/or bulbar dysfunction). Assessments will include medical history, physical exam, vital signs and bloodwork. MG assessments will also be conducted including the QMG and MG-ADL and patient reported outcome measures like the Myasthenia Gravis Quality of Life 15 item Revised (MGQoL15r) scale. Treatment will start in the hospital and once the patient is discharged, treatment will continue as an outpatient. Current medications and adverse events will also be reviewed and documented. Patients who undergo treatment with zilucoplan will be vaccinated against meningitis prior to starting the study drug and will continue with the recommended set of vaccines for 6 months. Antibiotics will be taken concurrently until patients are fully vaccinated.

The study aims to find a less invasive method to treat MG patients who are experiencing an exacerbation. Utilization of a subcutaneous medication with relatively rapid onset of action may provide a viable alternative to the current therapeutic approaches. If rapid complement inhibition were to prove efficacious in the treatment of acute exacerbations of gMG, this therapy would potentially obviate the need for transfer to tertiary care centers, avoid the potentially hazardous placement of a large bore central venous catheter for plasmapheresis, and potentially reduce hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient determined to have severe MG exacerbation (e.g. bulbar and/or respiratory symptoms requiring hospitalization, neck extension weakness)
* MGFA class II - IVb
* Male or female aged ≥18
* MG-ADL ≥6 in non-ocular domains
* Serology - AChR antibody positive (or historically available data)
* If female of child-bearing potential (i.e., not surgically sterile or post-menopausal defined as age > 51 years without menses for ≥ 2 years), negative serum pregnancy test at screening
* Women of child-bearing potential or men with sexual partners of childbearing potential must be willing to use an acceptable method of birth control for the duration of the study and for 40 days after the last dose of study drug therapy. Acceptable methods of birth control include abstinence, oral contraceptives, the contraceptive patch, intra-uterine device, the contraceptive ring, and or barrier contraception such as condoms with spermicide.
* Completed or updated meningococcal vaccination or initiated meningococcal vaccination with appropriate antibiotic prophylaxis according to current USPI and ACIP guidelines

Exclusion Criteria:

* History of meningococcal disease
* Participants requiring intubation prior to study start.
* Recent significant infections which could have caused exacerbation e.g. sepsis and wound infections
* Pregnancy or lactating
* Recent surgery (<4 weeks). Minor procedures/surgeries allowed at the discretion of the site principal investigator
* Current use or known failure of C5 inhibitors in the previous 3 months
* Initiation of plasma exchange or IVIG in the past 4 weeks
* Participation in concurrent clinical trial with a therapeutic medication
* Rituximab use in the previous 9 months
* Any clinically significant condition or illness, which, in the opinion of the PI, would pose a risk to the subject or might confound the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 2 in the Myasthenia Gravis - Activities of Daily Living (MG-ADL) score | From baseline to Week 2
  The MG-ADL is an assessment that measures MG symptom severity. There are 8 items measured on a scale of 0-3 with 0 being the least severe. The total of the 8 items represents the MG-ADL score. The score can range from 0 (least severe) to 24 (most severe).

SECONDARY OUTCOMES:
Change from baseline to week 12 in Myasthenia Gravis - Activities of Daily Living (MG-ADL) score | From baseline to week 12
  The MG-ADL is an assessment that measures MG symptom severity. There are 8 items measured on a scale of 0-3 with 0 being the least severe. The total of the 8 items represents the MG-ADL score. The score can range from 0 (least severe) to 24 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Freimer, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vu T, Meisel A, Mantegazza R, Annane D, Katsuno M, Aguzzi R, Enayetallah A, Beasley KN, Rampal N, Howard JF. Terminal Complement Inhibitor Ravulizumab in Generalized Myasthenia Gravis. NEJM Evid. 2022 May;1(5):EVIDoa2100066. doi: 10.1056/EVIDoa2100066. Epub 2022 Apr 26. PMID 38319212
- [Background] Howard JF Jr, Bresch S, Genge A, Hewamadduma C, Hinton J, Hussain Y, Juntas-Morales R, Kaminski HJ, Maniaol A, Mantegazza R, Masuda M, Sivakumar K, Smilowski M, Utsugisawa K, Vu T, Weiss MD, Zajda M, Boroojerdi B, Brock M, de la Borderie G, Duda PW, Lowcock R, Vanderkelen M, Leite MI; RAISE Study Team. Safety and efficacy of zilucoplan in patients with generalised myasthenia gravis (RAISE): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Neurol. 2023 May;22(5):395-406. doi: 10.1016/S1474-4422(23)00080-7. PMID 37059508
- [Background] Kusner LL, Kaminski HJ. The role of complement in experimental autoimmune myasthenia gravis. Ann N Y Acad Sci. 2012 Dec;1274(1):127-32. doi: 10.1111/j.1749-6632.2012.06783.x. PMID 23252907
- [Background] Kapoor M, Spillane J, Englezou C, Sarri-Gonzalez S, Bell R, Rossor A, Manji H, Reilly MM, Lunn MP, Carr A. Thromboembolic risk with IVIg: Incidence and risk factors in patients with inflammatory neuropathy. Neurology. 2020 Feb 11;94(6):e635-e638. doi: 10.1212/WNL.0000000000008742. Epub 2019 Dec 18. PMID 31852814
- [Background] Mandawat A, Kaminski HJ, Cutter G, Katirji B, Alshekhlee A. Comparative analysis of therapeutic options used for myasthenia gravis. Ann Neurol. 2010 Dec;68(6):797-805. doi: 10.1002/ana.22139. PMID 21061395
- [Background] Chang CC, Yeh JH, Chiu HC, Liu TC, Chen YM, Jhou MJ, Lu CJ. Assessing the length of hospital stay for patients with myasthenia gravis based on the data mining MARS approach. Front Neurol. 2023 Dec 14;14:1283214. doi: 10.3389/fneur.2023.1283214. eCollection 2023. PMID 38156090
- [Background] Sanders DB, Wolfe GI, Benatar M, Evoli A, Gilhus NE, Illa I, Kuntz N, Massey JM, Melms A, Murai H, Nicolle M, Palace J, Richman DP, Verschuuren J, Narayanaswami P. International consensus guidance for management of myasthenia gravis: Executive summary. Neurology. 2016 Jul 26;87(4):419-25. doi: 10.1212/WNL.0000000000002790. Epub 2016 Jun 29. PMID 27358333
- [Background] Wolfe GI, Kaminski HJ, Aban IB, Minisman G, Kuo HC, Marx A, Strobel P, Mazia C, Oger J, Cea JG, Heckmann JM, Evoli A, Nix W, Ciafaloni E, Antonini G, Witoonpanich R, King JO, Beydoun SR, Chalk CH, Barboi AC, Amato AA, Shaibani AI, Katirji B, Lecky BR, Buckley C, Vincent A, Dias-Tosta E, Yoshikawa H, Waddington-Cruz M, Pulley MT, Rivner MH, Kostera-Pruszczyk A, Pascuzzi RM, Jackson CE, Garcia Ramos GS, Verschuuren JJ, Massey JM, Kissel JT, Werneck LC, Benatar M, Barohn RJ, Tandan R, Mozaffar T, Conwit R, Odenkirchen J, Sonett JR, Jaretzki A 3rd, Newsom-Davis J, Cutter GR; MGTX Study Group. Randomized Trial of Thymectomy in Myasthenia Gravis. N Engl J Med. 2016 Aug 11;375(6):511-22. doi: 10.1056/NEJMoa1602489. PMID 27509100
- [Background] Ramizuddin MK. Review on: Myasthenia gravis and telithromycin-myasthenia crisis. IOSR J Dent Med Sci. 2014;13(7):67-97.
- [Background] Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016 Dec 29;375(26):2570-2581. doi: 10.1056/NEJMra1602678. No abstract available. PMID 28029925
- [Background] Howard JF Jr, Utsugisawa K, Benatar M, Murai H, Barohn RJ, Illa I, Jacob S, Vissing J, Burns TM, Kissel JT, Muppidi S, Nowak RJ, O'Brien F, Wang JJ, Mantegazza R; REGAIN Study Group. Safety and efficacy of eculizumab in anti-acetylcholine receptor antibody-positive refractory generalised myasthenia gravis (REGAIN): a phase 3, randomised, double-blind, placebo-controlled, multicentre study. Lancet Neurol. 2017 Dec;16(12):976-986. doi: 10.1016/S1474-4422(17)30369-1. Epub 2017 Oct 20. PMID 29066163
- [Background] Rodrigues E, Umeh E, Aishwarya, Navaratnarajah N, Cole A, Moy K. Incidence and prevalence of myasthenia gravis in the United States: A claims-based analysis. Muscle Nerve. 2024 Feb;69(2):166-171. doi: 10.1002/mus.28006. Epub 2023 Dec 1. PMID 38040629
- See also: Zilbrysq Package Insert — https://www.ucb-usa.com/zilbrysq-prescribing-information.pdf
- See also: Advisory Committee on Immunization Practices (ACIP) Vaccine Recommendations — https://www.cdc.gov/mmwr/volumes/73/wr/pdfs/mm7349a3-H.pdf